CLINICAL TRIAL: NCT05703087
Title: The Effect of Positive Cueing in the Information Video for Patients Undergoing Total Knee Arthroplasty: a Feasibility Study for a Randomized Controlled Trial.
Brief Title: Positive Cueing in Knee Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Rudolf W Poolman, MD PhD, Clinical Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WO 21.122
Record Dates: First submitted 2023-01-08; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Psychological Stress; Mental Stress
MeSH Terms: conditions — Osteoarthritis, Knee; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: A single-center feasibility study. We compared the use of positive cueing in the information video before a primary total knee arthorplasty (TKA) with the standard information video.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard information video before primary total knee arthroplasty (No Intervention): Information video (about procedure, complications, rehabilitation) shown to the participants before TKA in the OLVG.
- Positive cueing in the information video before a primary total knee arthroplasty (Experimental): The information video was adapted from the existing standard information video used in OLVG. The concept of positive cueing was applied to the standard video by an expert team including a psychiatrist and clinical psychologist. Illustrations which were incomprehensible or with negative associations were removed.
  Four rules were followed to use positive cueing:
  1. make patients aware that they are able to influence their own recovery process,
  2. be descriptive in explanations; objectively describe the performed procedure, name equivalent, not negatively charged feelings,
  3. explain why specific steps and actions during the procedure are performed, so the patients understand what is going to happen,
  4. do not use medical langue, but use accessible, understandable language instead.
  Interventions: Behavioral: Positive cueing in the information video before a primary TKA

INTERVENTIONS:
Behavioral: Positive cueing in the information video before a primary TKA — Two weeks before the surgery, in the outpatient clinic (during their preoperative appointment), the pre-surgery information video was shown to the patients. Patients were randomly allocated to either the positive cueing group (intervention) or the standard care group (control) with Castor EDC (14) using a variable block randomization model. Patients did not know whether they watched the adapted video or the standard video.
  Arms: Positive cueing in the information video before a primary total knee arthroplasty

SUMMARY:
To the knowledge of the investigators, the feasibility of an RCT assessing the use of positive cueing in an information video for patients undergoing primary TKA is currently unclear.

The investigators conducted a feasibility study with the primary objective to assess the acceptability of the randomized controlled trial (RCT) procedure for participating patients. The secondary objective was to evaluate the rate of recruitment, the comprehensibility (do patients understand what is expected of them during the trial) and if there were any adjustments necessary to the design of the study. The outcome of the current feasibility study will be used to determine whether adjustments are required to the design of the RCT before we proceed.

DETAILED DESCRIPTION:
Even though total knee arthroplasty (TKA) is a cost-effective treatment, 10 - 34% of the patients report pain and discomfort up to two years after the procedure. Preoperative symptoms of anxiety and/or depression (which is present in approximately 10 - 58.6% of TKA patients seem to be related to poor pain coping techniques, which can lead to higher levels of pain up to two years after surgery. Our previous systematic review showed that a reduction of preoperative symptoms of anxiety and depression may lead to a reduction of postoperative pain after TKA.

In radiology, anesthesiology, and pediatric departments multiple studies have been performed on reducing the perception of pain with the use of language and hypnosis. This led to the concept of positive cueing. With positive cueing, general language without negative suggestions is used in provided information and instructions about the management of potential discomfort. Correct use of positive cueing has been shown to improve patients' satisfaction and to decrease need for additional treatments (such as blood transfusion) after several medical procedures, whereas use of negative language (warning patients for pain or negative experiences) seems to result in higher pain and anxiety scores.

Before TKA, patients are informed about the procedure and the risk of complications. Positive cueing might positively influence perioperative anxiety symptoms and subsequently improve pain after TKA. The investigators plan to conduct a randomized controlled trial (RCT) to address the question whether the use of positive cueing in the information video for patients undergoing a primary TKA, compared to the standard care video, will reduce the level of preoperative symptoms of anxiety and improve pain coping styles.

To the knowledge of the reviewers, no previous studies addressed this topic. Hence, the feasibility of an RCT assessing the use of positive cueing in an information video for patients undergoing primary TKA is currently unclear. As such, this feasibility study was conducted with the primary objective to assess the acceptability of the RCT procedure for participating patients. Secondly, the rate of recruitment, the comprehensibility (do patients understand what is expected of them during the trial) and if there were any adjustments necessary to the design of the study were evaluated. The outcome of the current feasibility study will be used to determine whether adjustments are required to the design of the RCT before the investigators proceed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* end-stage knee osteoarthritis for which participants were scheduled for a TKA
* sufficient Dutch languages skills to understand the information video
* able to fill out the questionnaires.

Exclusion Criteria:

* not receiving TKA for osteoarthritis of the knee
* not sufficient Dutch languages skills to understand the information video
* not able to fill out the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome measure: acceptibility. | During the preoperative outpatient clinic visit two weeks before surgery. Directly after watching the video's and completing questionnaires.
  The primary feasibility outcome score was the acceptability to participate, assessed with a developed questionnaire.
  The investigators conducted a questionnaire about the experience of the participants with a Likart scale 1 - 5, existing of 4 questions. A total score of 12 or higher was interpreted as acceptable since the patient seemed have a positive experience according to the questionnaire. As part of the primary outcome measure (acceptibility), we monitored the time it took a patient to participate in the study. The study should not take more than one hour to be acceptable.

SECONDARY OUTCOMES:
Feasibility outcome measure: rate of recruitment | The number of the patients on the waiting list for total knee arthroplasty and the included patients were assessed two weeks before surgery, during the outpatient clinic visit.
  We determined the rate of recruitment by dividing the number of patients included in this study by the number of patients waiting for total knee arthroplasty meeting all inclusion criteria who were scheduled to be seen on the preoperative outpatient clinic appointment.
Feasibility outcome measure: comprehensibility | During the preoperative outpatient clinic visit two weeks before surgery. Directly after watching the video's and completing questionnaires.
  Do patients understand what is expected of them during the trial. We analyzed comprehensibility for the patients with a developed questionnaire with a cut off point < 9 and by assessing the rate of completion of the questionnaires (number of questions completed). Specific items that were consistently missing from the questionnaires and were not filled out by the patients were noted. Also, patients received one question about whether they thought the information in the video was easy to understand, cut off point < 3.
Feasibility outcome measure:patients' feedback to the current protocol. | During the preoperative outpatient clinic visit two weeks before surgery. Directly after watching the video's and completing questionnaires.
  After finishing the questionnaire we asked two feedback questions regarding the protocol:
  1. what patients thought of participating in the study, and
  2. whether they had suggestions to improve the study process. The feedback from the patients were transcribed and similar answers were categorized.

CONTACTS AND LOCATIONS:
Locations (1):
- LUMC, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No